CLINICAL TRIAL: NCT00935883
Title: Eculizumab for the Treatment of Non-Exudative Age-Related Macular Degeneration: An Exploratory Study to Evaluate the Effects of C5 Inhibition on Drusen and Geographic Atrophy
Brief Title: Complement Inhibition With Eculizumab for the Treatment of Non-Exudative Macular Degeneration (AMD)
Acronym: COMPLETE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philip J. Rosenfeld, MD, PhD (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Philip J. Rosenfeld, MD, PhD, Professor of Ophthalmology, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20090055
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age Related macular Degeneration; Macular Degeneration; Drusen; Geographic atrophy; Eculizumab; Soliris
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — eculizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Randomized patients in the drusen or the GA cohort will receive placebo saline infusions as a comparator
  Interventions: Drug: Saline
- Eculizumab (Active Comparator): Randomized patients in the drusen or the GA cohort will receive active treatment with eculizumab
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Induction Period: patient will receive eculizumab 600 mg or 900 mg via IV infusion over approximately 30 minutes once a week (7 ± 2 days) for 4 weeks followed by 900 mg or 1200 mg eculizumab for the fifth dose 7 days later (7 ± 2 days).
  Maintenance Period: patient will receive eculizumab 900 mg or 1200 mg via IV infusion over approximately 30 minutes every 2 weeks (14 ± 2 days) until week 24.
  Observation period: patient will then be observed for 6 months off treatment with follow-up visits scheduled for 9 months and 12 months.
  Other Names: Soliris
  Arms: Eculizumab
Drug: Saline — Induction Period: patient will receive saline via IV infusion over approximately 30 minutes once a week (7 ± 2 days) for 4 weeks followed by saline for the fifth dose 7 days later (7 ± 2 days).
  Maintenance Period: patient will receive saline via IV infusion over approximately 30 minutes every 2 weeks (14 ± 2 days) until week 24.
  Observation period: patient will then be observed for 6 months off treatment with follow-up visits scheduled for 9 months and 12 months.
  Other Names: PBS
  Arms: Saline

SUMMARY:
To evaluate the safety and efficacy of eculizumab for the treatment of dry AMD as evaluated by the change in drusen volume and area of geographic atrophy.

DETAILED DESCRIPTION:
This is a randomized, double-arm, double-masked study designed to evaluate the safety and efficacy of eculizumab for the treatment of patients with dry AMD. There are three stages in the study: the screening period, the treatment period, and the follow-up period.During the screening period patients will be evaluated for eligibility. Eligible patients will receive either eculizumab or placebo for 24 weeks.

A total of 60 patients will be enrolled and divided equally between the drusen cohort and the GA cohort. A 2:1 randomization will result in 20 patients in each cohort receiving eculizumab while 10 patients receive placebo.

The treatment period will begin two weeks after administration of the meningococcal vaccine. During the treatment period, patients will receive eculizumab or placebo over a period of approximately 26 weeks. Patient will treatment according to the following regimen:

Induction Period: patient will receive eculizumab 600 mg or 900 mg via IV infusion over approximately 30 minutes once a week (7 ± 2 days) for 4 weeks followed by 900 mg eculizumab for the fifth dose 7 days later (7 ± 2 days).

Maintenance Period: patient will receive eculizumab 900 mg or 1200 mg via IV infusion over approximately 30 minutes every 2 weeks (14 ± 2 days).

After the final scheduled dose of eculizumab or Placebo at week 24, patients will return for follow-up exam 2 weeks, 3 months, and 6 months after the final dose.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* In the study eye(s), the presence of non-exudative AMD documented by fundus photography, autofluorescence, fluorescein angiography, and spectral domain OCT.
* Visual acuity of 20/63 or better (BCVA score of at least 59 letters) as measured on an ETDRS chart.
* Able and willing to comply with study procedures.

Exclusion Criteria:

* Visual acuity worse than 20/63
* Any history of choroidal neovascularization in the study eye
* Unresolved meningococcal disease.
* Confounding ocular conditions such as amblyopia; aphakia; myopia requiring >6 diopters of correction; pigment epithelial detachment; uncontrolled glaucoma (intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication); steroid-induced ocular hypertension; retinal inflammatory disease; central serous choroidopathy; prior or current retinal detachment; macular edema; cystic lesion (individual cysts or cystoid macular edema); ocular herpes simplex virus; severe non-proliferative or worse diabetic retinopathy; anterior ischemic optic neuropathy; RPE tear involving the macula; pseudovitelliform macular degeneration; vitreo-retinal traction maculopathy; vitreous hemorrhage, history of or current rhegmatogenous retinal detachment or macular hole; uveitis; diffuse choroidal atrophy; optic atrophy (as evidenced by pallor); intraocular inflammation; ocular or periocular infection; moderate or worse dry eye syndrome; clinically significant cataract or opacification of the posterior capsule which, in the Investigator's opinion, would progress during the course of the study and could affect central vision; other ocular conditions that the Investigator believes may be a confounding factor in this study
* Refusal to be vaccinated against Neisseria meningitides or an active Neisseria meningitides infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Rosenfeld, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

REFERENCES:
- [Result] Yehoshua Z, de Amorim Garcia Filho CA, Nunes RP, Gregori G, Penha FM, Moshfeghi AA, Zhang K, Sadda S, Feuer W, Rosenfeld PJ. Systemic complement inhibition with eculizumab for geographic atrophy in age-related macular degeneration: the COMPLETE study. Ophthalmology. 2014 Mar;121(3):693-701. doi: 10.1016/j.ophtha.2013.09.044. Epub 2013 Nov 26. PMID 24289920
- [Result] Garcia Filho CA, Yehoshua Z, Gregori G, Nunes RP, Penha FM, Moshfeghi AA, Zhang K, Feuer W, Rosenfeld PJ. Change in drusen volume as a novel clinical trial endpoint for the study of complement inhibition in age-related macular degeneration. Ophthalmic Surg Lasers Imaging Retina. 2014 Jan-Feb;45(1):18-31. doi: 10.3928/23258160-20131217-01. PMID 24354307
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- [Derived] Stetson PF, Yehoshua Z, Garcia Filho CA, Portella Nunes R, Gregori G, Rosenfeld PJ. OCT minimum intensity as a predictor of geographic atrophy enlargement. Invest Ophthalmol Vis Sci. 2014 Feb 10;55(2):792-800. doi: 10.1167/iovs.13-13199. PMID 24408973

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: Randomized patients in the drusen or the GA cohort will receive placebo saline infusions as a comparator
  Saline: Induction Period: patient will receive saline via IV infusion over approximately 30 minutes once a week (7 ± 2 days) for 4 weeks followed by saline for the fifth dose 7 days later (7 ± 2 days).
  Maintenance Period: patient will receive saline via IV infusion over approximately 30 minutes every 2 weeks (14 ± 2 days) until week 24.
  Observation period: patient will then be observed for 6 months off treatment with follow-up visits scheduled for 9 months and 12 months.
- Eculizumab: Randomized patients in the drusen or the GA cohort will receive active treatment with eculizumab
  Eculizumab: Induction Period: patient will receive eculizumab 600 mg or 900 mg via IV infusion over approximately 30 minutes once a week (7 ± 2 days) for 4 weeks followed by 900 mg or 1200 mg eculizumab for the fifth dose 7 days later (7 ± 2 days).
  Maintenance Period: patient will receive eculizumab 900 mg or 1200 mg via IV infusion over approximately 30 minutes every 2 weeks (14 ± 2 days) until week 24.
  Observation period: patient will then be observed for 6 months off treatment with follow-up visits scheduled for 9 months and 12 months.
Period: Treatment Period
Arm/Group | Saline | Eculizumab
Started | 20 | 40
Completed | 19 | 38
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Follow-Up Period
Arm/Group | Saline | Eculizumab
Started | 19 | 38
Completed | 19 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Eculizumab | Total
Number analyzed (Participants) | 20 | 40 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 17 | 34 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (8.64) | 75.1 (8.0) | 75.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 29
  Male | 10 | 21 | 31
Region of Enrollment [Number; unit: participants]
  United States | 20 | 40 | 60

OUTCOME MEASURES:

1. Primary Outcome: Growth of Geographic Atrophy
Time Frame: 6 months
Population: Geographic Atrophy Cohort included 10 eyes randomized to saline and 20 eyes randomized to Eculizumab
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Saline | Eculizumab
Number analyzed (Participants) | 10 | 20
millimeters | 0.18 (0.15) | 0.19 (0.12)

2. Secondary Outcome: Change in Visual Acuity for Drusen Group
Description: Visual function was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better functioning. Maximum score would be 100 letters read and minimum would be count fingers, hand motion and light perception if there were no letters read on the chart.
Time Frame: Baseline/ 6 Months
Population: Drusen Cohort included 10 eyes randomized to saline and 20 eyes randomized to Eculizumab
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Saline | Eculizumab
Number analyzed (Participants) | 10 | 20
letters | 4.0 (7.0) | 2.4 (3.9)

3. Primary Outcome: Decrease in Drusen Volume
Time Frame: 6 Months
Population: Drusen Cohort included 10 eyes randomized to saline and 20 eyes randomized to Eculizumab
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Saline | Eculizumab
Number analyzed (Participants) | 10 | 20
mm^3 | 0.12 (0.08) | 0.15 (0.17)

4. Secondary Outcome: Change in Visual Acuity for Geographic Atrophy Group
Description: as for outcome 2
Time Frame: Baseline/ 6 Months
Population: Geographic Atrophy Cohort included 10 eyes randomized to saline and 20 eyes randomized to Eculizumab
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Saline | Eculizumab
Number analyzed (Participants) | 10 | 20
letters | -2.6 (7.2) | 2.5 (4.1)

ADVERSE EVENTS:
Arm/Group | Saline | Eculizumab
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/40
Other Adverse Events (participants affected / at risk) | 1/20 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=20) | Eculizumab (N=40)
chest pains (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No